CLINICAL TRIAL: NCT05428553
Title: Endoscopic Cold Snare Polypectomy Versus Endoscopic Mucosal Resection of Superficial Non-ampullary Duodenal Tumors (SNADTs) (>6mm, Sessile) - A Prospective Multicenter Historically Controlled Trial
Brief Title: CSP vs EMR for >6mm Superficial Non-ampullary Duodenal Tumors
Acronym: CSP; EMR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShanghaiZhongshanEndoscopy1
Record Dates: First submitted 2022-03-20; First posted 2022-06-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-03

CONDITIONS: Duodenal Tumor
MeSH Terms: conditions — Duodenal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSP/p-CSP (Experimental): Prospective allocation
  Interventions: Procedure: Endoscopic resection: CSP/p-CSP
- EMR/EPMR (Active Comparator): Historical control
  Interventions: Procedure: Endoscopic resection: EMR/EPMR

INTERVENTIONS:
Procedure: Endoscopic resection: CSP/p-CSP — Patients in the experimental arm will be assigned to receive CSP/p-CSP.
  Arms: CSP/p-CSP
Procedure: Endoscopic resection: EMR/EPMR — Patients in the historical control arm have already finished EMR/EPMR
  Arms: EMR/EPMR

SUMMARY:
There is currently no reliable evidence on the safety of CSP (cold snare polypectomy) / p-CSP (piecemeal CSP) for SNADT greater than 6mm.In this prospective historical controlled study, we intend to test the role of CSP / p-CSP in the treatment of pedicle less snadt greater than 6mm compared with EMR (endoscopic mucosal resection) / EPMR (endoscopic piecemeal mucosal resection).

DETAILED DESCRIPTION:
Due to the possibility of malignant transformation of duodenal adenomatous lesions, endoscopic resection is recommended as far as possible. The European Society of endoscopy guidelines recommend cold snare polypectomy for superficial non ampullary duodenal tumors (SNADT) less than 6mm in diameter, while EMR (endoscopic mucosal resection) is recommended as a first-line endoscopic resection for other larger lesions. ESD (endoscopic submucosal dissection) is not considered as the standard treatment of duodenum due to its difficult operation and high complication rate.

In recent years, CSP (cold snare polypectomy) has been widely used in the colon. CSP is a safe alternative method of directly removing polyps with snare without electrifying. Reducing electrocoagulation can reduce the damage of peripheral blood vessels and intestinal wall, leading to decreased risk of delayed bleeding and perforation. CSP has gradually replaced EMR in the resection of colorectal lesions of appropriate size.

So far, there is no reliable evidence on the safety of CSP / p-CSP (piecemeal CSP) for SNADT greater than 6mm.In this prospective historical controlled study, we intend to test the role of CSP / p-CSP in the treatment of pedicle less snadt greater than 6mm compared with EMR / EPMR (endoscopic piecemeal mucosal resection).

ELIGIBILITY:
Inclusion Criteria:

Experimental arm: CSP/p-CSP

1. Patients of age 18-75 years.
2. Lesion located in the duodenum.
3. Superficial non-ampullary duodenal tumors (SNADTs) (>6mm, Sessile).
4. Written informed consent.
5. Benign adenomatous surface features (Kudo III / IV, JNET(Japan NBI (narrow-band imaging) Expert Team) 2a).

Control arm: EMR/EPMR

1. Patients of age 18-75 years.
2. Lesion located in the duodenum.
3. Superficial non-ampullary duodenal tumors (SNADTs) (>6mm, Sessile).
4. Benign adenomatous surface features (Kudo III / IV, JNET 2a).
5. Received EMR/EPMR already.
6. Provided written informed consent for use of clinical information.

Exclusion Criteria:

Experimental arm: CSP/p-CSP

1. Absence of proper suspension of the anticoagulant/antiplatelet therapy prior to procedure according to usual pre-procedure recommendations according to the guidelines, or presence of coagulation disorder （PLT (platelet)<50×10^9 / L or INR (international normalized ratio)≥1.5) at the time of EMR/EPMR.
2. History of surgery in the stomach or duodenum (endoscopic surgery not included), or receiving chemotherapy/radiotherapy at the time of EMR/EPMR.
3. Pregnant or breast feeding at the time of EMR/EPMR.
4. Lesions involving the ampullary area.
5. Endoscopic features suggestive of submucosal invasion (Kudo Vi/n, JNET 2b / 3).
6. Scar of previous endoscopic procedures within 10mm around the lesion.

Control arm: EMR/EPMR

1. Absence of proper suspension of the anticoagulant/antiplatelet therapy prior to procedure according to usual pre-procedure recommendations according to the guidelines, or presence of coagulation disorder （PLT<50×10^9 / L or INR≥1.5)；.
2. History of surgery in the stomach or duodenum (endoscopic surgery not included), or receiving chemotherapy/radiotherapy.
3. Pregnant or breast feeding.
4. Lesions involving the ampullary area.
5. Endoscopic features suggestive of submucosal invasion (Kudo Vi/n, JNET 2b / 3).
6. Scar of previous endoscopic procedures within 10mm around the lesion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 2 weeks
  iIntraoperative and postoperative adverse events; through medical records and telephone follow up

SECONDARY OUTCOMES:
Postoperative adverse events | 2 weeks
  postoperative adverse events; through medical records and telephone follow up
Clinically significant delayed bleeding | 2 weeks
  Leading to emergency room visit, readmission, or intervention
Delayed perforation | 2 weeks
  Image confirmed
Clinically significant intra-procedural bleeding Intraoperative adverse events Delayed perforation | intra-procedural
  Not responsive to water flushing and clips are needed
Intraoperative deep mural injury | intra-procedural
  stage III/IV/V
En bloc resection | intra-procedural
  specimen resected in one piece
Procedure duration | intra-procedural
  the entire duration of the procedure, not including ascending of the scope and looking for the lesions
Recurrence after 6 months | 6 months
  confirmed by colonoscopy

OTHER OUTCOMES:
Cost | 2 weeks
  total cost of hospitalization
Number of treatment after technical failure | 6 months
  through medical records and telephone follow up
Number of clips | intra-procedural
  number of clips used to close the wound

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Hong Zhou, MD,PhD, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Original data could be shared at request by email after publication
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: The data will be available after publication of the study
Access Criteria: The shared data could be available by contacting Dr. Xin-Yang Liu at shmulxy@163.com.